CLINICAL TRIAL: NCT02963337
Title: Pain Relief and Progress of Labour With Remifentanil Patient-controlled Analgesia Versus Combined Spinal-epidural Analgesia in Multiparous Women: a Prospective Observational Study
Brief Title: Remifentanil vs. Combined Spinal-epidural Analgesia for Labor Analgesia and Progress of Labor in Multiparous
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tatjana Stopar Pintaric, Associate Professor, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 2104
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Labor Pain; Labor; Prolonged, Second Stage; Labor; Prolonged, First Stage
Keywords: remifentanil; combined spinal-epidural analgesia; multiparous
MeSH Terms: conditions — Labor Pain | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- remifentanil PCA: The patients in the remifentanil group will receive remifentanil hydrochloride (Ultiva, GlaxoSmithKline, Oslo, Norway) diluted in physiologic saline to a concentration of 40µg/ml and administered using PCA pump with a bolus duration of 20 sec. A stepwise bolus doses from 15 to 30 µg, maximum 40 per 2 min will be applied with no background infusion.
  Interventions: Drug: remifentanil
- Combined spinal-epidural analgesia PCA: A 27-gauge needle will be placed via the shaft of the epidural needle inserted at the L2-3/L3-4 inter-space by the investigator. After confirming the CSF, 2,5 mg of bupivacaine with 20 µg of fentanyl will be injected. That will be followed by the placement of a 20-gauge multi-hole catheter into the epidural space which will be connected to the PCA pump with a possibility of injecting 6-10 ml 0,1% bupivacaine with 2 µg of fentanyl/ml every 20 min with no background infusion.
  Interventions: Drug: combined spinal-epidural analgesia

INTERVENTIONS:
Drug: remifentanil — Remifentanil PCA will be used to deliver intravenous drug boluses from 20 to 40 micrograms per 2 min lockout interval.
  Other Names: ULTIVA
  Groups: remifentanil PCA
Drug: combined spinal-epidural analgesia — Patient controlled epidural analgesia will be used to deliver epidural boluses of 6-10 ml of 0,1% bupivacaine with 2 micrograms of fentanyl per ml per 15 min lockout interval.
  Other Names: bupivacaine epidurally
  Groups: Combined spinal-epidural analgesia PCA

SUMMARY:
Remifentanil may be an ideal drug for labor analgesia due to its pharmacodynamic and pharmacokinetic profile. As compared to epidural analgesia, it demonstrated satisfactory for pain relief at the beginning of labour with a gradual elevation of pain scores as labour progresses. However, fast onset and limited time efficacy may render it useful in multiparous with a faster labor progression, thus even making it an alternative to single-shot spinal analgesia.

DETAILED DESCRIPTION:
Introduction:

Neuraxial analgesia is considered the most effective method of pain relief during labor. When unavailable, contraindicated, refused by parturient or discouraged by midwife/obstetrician, alternative methods of analgesia are required which should to be effective, without major side effects and flexible enough to adapt to variable analgesic requirements during labor.

Remifentanil may be an ideal drug for labor analgesia due to its pharmacodynamic and pharmacokinetic profile. It is an ultra-short-acting µ1-opioid receptor agonist, rapidly metabolized by plasma and tissue esterases. It has onset time of 30 to 60 seconds and a peak effect at 2,5 min. It rapidly crosses the placenta and it is quickly metabolized by the fetus. Several studies which compared remifentanil patient controlled analgesia (PCA) with epidural analgesia in nulliparous patients or parturient of mixed parity have demonstrated a lower analgesic efficacy of remifentanil. Remifentanil, as compared to epidural analgesia, showed a satisfactory for pain relief only at the beginning of labor with a gradual elevation of pain scores as labor progressed. However, the fast onset and limited time efficacy may render it useful in multiparous with a faster labor progression, thus even making it an alternative to single-shot spinal analgesia.

The anaesthetic technique may also affect the progress of labor. A combined spinal-epidural analgesia (CSEA) has been demonstrated to be associated with a greater cervical dilation relative to conventional epidural analgesia in nulliparous patients. There are no data on labour progression difference as compared to remifentanil PCA in multiparous.

We therefore conduct the study in multiparous patients to compare remifentanil PCA and CSEA with respect to pain relief and the progress of labor.

Methods:

Approval for this observational trial was obtained by Republic of Slovenia National Ethical Committee (kme.mz@gov.si). Only multiparous fulfilling inclusion criteria will be recruited. The parturient requesting remifentanil analgesia will receive remifentanil hydrochloride (Ultiva, GlaxoSmithKline, Oslo, Norway) according to the standard operative protocol. Bolus doses will be adjusted by anesthesia staff on patient request and side effects (level of sedation <3 according to Ramsey scale (scale1-5: 1= alert, 2 = slightly drowsy, 4 = very drowsy, 5 = unarousable), respiratory rate (RR)>8 breaths per min, oxygen saturation (SaO2) >94%, systolic blood pressure (SBP) > 90 mmHg, heart rate (HR) > 50/min and acceptable overall clinical assessment performed by the investigator). Women using remifentanil will have one-to-one midwifery care. All midwives will be familiar with the protocol and have already received training in this mode of analgesia. Respiratory monitoring will be performed throughout the labor only in the remifentanil group using a Capno stream capnograph with an oral-nasal cannula, sampling from both the nose and mouth. Supplemental oxygen (2L/min via nasal catheter) will be given in all patients. Respiratory monitoring will record continuous waveform end-tidal carbon dioxide (ETCO2), SBP, SaO2 and maternal HR. The audible alarms will be activated with SaO2<94%, RR<8/min and apnea longer than 20 sec which triggered a staged intervention starting with a verbal command and/or light tap on the parturient arm.

CSEA will be provided on parturient request according to the standard operative protocol. Fetal heart rate (FHR) will be monitored to ensure neonatal safety using cardiotocography.

Data acquisition and retrieval:

Demographic and medical data will be obtained from personal interviews before analgesia initiation and throughout the labor.

Maternal pain will be evaluated using a 11-point verbal numerical rating scale (NRS), where 0 is no pain and 10 is the worst imaginable pain. NRS pain scores will be recorded immediately before starting PCA (baseline), then every 15 min during the first hour and every 30 min thereafter.

Patient satisfaction with pain relief will be evaluated every 30 minutes after analgesia administration and within 24 hours after delivery using a five-point categorical scale (1=very good, 2=good, 3=moderate, 4=poor, 5=very poor). At the same time, each parturient will be asked if she would choose the same technique for the next delivery and/or recommend the same technique to somebody else.

Non-invasive SBP, maternal HR, SaO2 and sedation score will be recorded before analgesia and every 30 min thereafter. The respiratory monitor data will be recorded and adverse respiratory events (SaO2<94%, RR<8/min and apnea>20 sec) counted for each woman.

The number of epidural boluses as well as the total dose of remifentanil will be registered automatically in the PCA pump and recorded for each patient. Maternal requests for additional analgesia will be manually recorded.

Data concerning nausea, vomiting and itching will also be collected.

Oral temperature will be measured both at the onset of analgesia and within 1 hour of delivery.

Data on labor progress (first and second stage labor duration, mean cervical dilation rate) and outcome will be recorded for each patient, including the use and maximum dose of oxytocin administered, and mode of delivery (spintaneus vaginal, instrumental vaginal, caesarean section). Cervical dilation will be assessed by the midwife, and all changes recorded till delivery. The time from onset of analgesia until 10-cm cervical dilation will be defined as the first stage of labor, while the second stage will be defined as the interval between full cervical dilation and delivery of the neonate. The mean cervical dilation rate will be defined as 10 minus last cervical examination before analgesia divided by time between examinations.

After delivery, Apgar score at 1 and 5 min,and umbilical artery pH and base excess will be abstracted from the medical records.

Sample size was calculated based on the primary outcome of pain relief during remifentanil and CSE analgesia in multiparous measured on an 11 point scale raging from 0 to 10. If the true difference between the two studied groups is 1 (on 11 point scale with estimated standard deviation of 2,2), we will need to study 77 subjects in each group to be able to reject the null hypothesis that the population means of the two groups are not equal with probability (power) 0,8. The Type I error probability associated with this test of this null hypothesis is 0,05.

ELIGIBILITY:
Inclusion Criteria:

* patients' request for pain relief
* ASA physical status 1-3
* uncomplicated singleton pregnancy with cefalic presentation
* gestation age > 37 weeks
* regular uterine contractions
* cervical dilation 2-5 cm
* anticipated vaginal delivery
* fetus without suspected abnormality and normal CTG

Exclusion Criteria:

* contraindications for remifentanil usage
* contraindications for CSE

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Multiparous
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Pain relief with remifentanil or CSE in multiparous women | two years
  Reduction in visual analog scoring after institution of the respective pain treatments

SECONDARY OUTCOMES:
Patient satisfaction with pain relief | two years
  Patient satisfaction with pain relief will be evaluated every 30 minutes after analgesia administration and within 24 hours after delivery using a five-point categorical scale (5=very good, 4=good, 3=moderate, 2=poor, 1=very poor). At the same time, each parturient will be asked if she would choose the same technique for the next delivery and/or recommend the same technique to somebody else.
Duration of first and second stage of labor | one year
  The time from onset of analgesia until 10-cm cervical dilation will be defined as the first stage of labor, while the second stage will be defined as the interval between full cervical dilation and delivery of the neonate. The mean cervical dilation rate will be defined as 10 minus last cervical examination before analgesia divided by time between examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Novak Jankovic, Professor, Study Chair — University Medical Centre
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Douma MR, Middeldorp JM, Verwey RA, Dahan A, Stienstra R. A randomised comparison of intravenous remifentanil patient-controlled analgesia with epidural ropivacaine/sufentanil during labour. Int J Obstet Anesth. 2011 Apr;20(2):118-23. doi: 10.1016/j.ijoa.2010.11.009. Epub 2011 Mar 3. PMID 21376564
- [Derived] Blajic I, Zagar T, Semrl N, Umek N, Lucovnik M, Stopar Pintaric T. Analgesic efficacy of remifentanil patient-controlled analgesia versus combined spinal-epidural technique in multiparous women during labour. Ginekol Pol. 2021;92(11):797-803. doi: 10.5603/GP.a2021.0053. Epub 2021 Apr 29. PMID 33914329